CLINICAL TRIAL: NCT00732017
Title: Effects Of High Voltage Pulsed Current On Ankle Post-Traumatic Injuries
Brief Title: Effects Of High Voltage Pulsed Current On Post-Traumatic Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Industrial de Santander (Other)
Responsible Party: Tania de Fátima Salvini, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5612
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Ankle Sprain
Keywords: Sprain; Electric stimulation; Physical trauma; Inflammation
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains; Wounds and Injuries; Inflammation | interventions — Electric Stimulation; Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HVPC- (Experimental): This group received standard physical therapy treatment and HVPC with negative polarity.
  Interventions: Device: high voltage pulse stimulation with negative polarity
- CG (Active Comparator): The control group received only standard physical therapy treatment.
  Interventions: Other: standard physical therapy treatment
- HVPC+ (Experimental): This group received standard physical therapy treatment and HVPC using active electrodes with positive polarity.
  Interventions: Device: Standard physical therapy and HVPC with positive polarity

INTERVENTIONS:
Device: Standard physical therapy and HVPC with positive polarity — A high voltage stimulator with positive polarity was used with a direct pulsed monophasic current, double peak, 5 and 8micros duration and separated by a pulsate interval of 75micros and monopolar application with a dispersive electrode in the lumbar region and two transarticular active electrodes. The intensity of the current was under motor level, that is, just before a visible motor response could be observed. The frequency used was 120pps, in a continuous mode and was applied once a day with thirty-minute duration.
  Other Names: electrical stimulation; electrical current
  Arms: HVPC+
Device: high voltage pulse stimulation with negative polarity — A high voltage stimulator with negative polarity was used with a direct pulsed monophasic current, double peak, 5 and 8micros duration and separated by a pulsate interval of 75micros and monopolar application with a dispersive electrode in the lumbar region and two transarticular active electrodes. The intensity of the current was under motor level, that is, just before a visible motor response could be observed. The frequency used was 120pps, in a continuous mode and was applied once a day with thirty-minute duration.
  Other Names: electrical stimulation; electrical current
  Arms: HVPC-
Other: standard physical therapy treatment — * Initial phase: Application of crushed ice on the ankle for 20 minutes. The subject performed isometric and active exercises of the ankle in all freedom degrees, with no weight bearing.
  * Intermediate phase: Application of cryotherapy continued and once mobility was completed and painless, progressive use of weight and reeducation of the walking pattern were initiated. Then, exercises with manual resistance of muscles of ankle and balance in stable surfaces were done.
  * Advanced phase: Balance exercises on unstable surfaces as well as strengthening ankle muscles with proprioceptive neuromuscular facilitation techniques and elastic band were performed. At the end, the patient did activities like trotting in S or Z and jumping in all directions.
  Other Names: standard care
  Arms: CG

SUMMARY:
The investigators hypothesis is that HVPC with negative polarity diminishes local post-traumatic edema in ankle sprains. Therefore, the objective of this study was to analyze the effect of HVPC on edema secondary to ankle sprains in humans.

DETAILED DESCRIPTION:
Most studies have investigated the effects of HVPC on edema in animals and only one in humans was identified. The studies had showed that HVPC had some advantages for controlling edema in animals but there are not yet conclusive results on the effect of this intervention in humans.For this reason, we proposed a randomized controlled double-blinded clinical trial with three groups of intervention. In our study compared the effects of standard physical therapy treatment with the HVPC with negative and positive polarity.

ELIGIBILITY:
Inclusion Criteria:

* Ankle post traumatic edema secondary to a sprain
* Sprain with evolution between 2 and 96 hours
* Sprain positive to anterior drawer test or lateral inclination mobilizations.

Exclusion Criteria:

* Subjects with grade III sprains that required surgical management
* Edema secondary to systemic illness
* Muscular dystrophy or atrophy
* Injuries, open or infected zones
* People taking anti-inflammatory medication or using empirical treatment as tractions, strong massages or manual.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-02; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Pain with the visual analogue scale. | The pain was measured before and at the end of the treatment.

SECONDARY OUTCOMES:
Range of movement (ROM) of plantar and dorsal flexion, inversion and eversion were measured with a goniometer. | The ROM was measured before and at the end of the treatment.
Edema was assessed with measures of ankle girth and volume. | The edema was measured before and at the end of the treatment.
Some descriptive variables of gait such as step and stride length, and the gait speed. | The variables of gait were measured before and at the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Sandoval Ortiz, M.Sc in P.T., Principal Investigator — Industrial University of Santander; Liliana Carolina Ramirez Ramirez, P.T., Principal Investigator — Industrial University of Santander; Diana Marina Camargo Lemos, M.Sc. Epid., Study Chair — Industrial University of Santander; Tania De Fatima Salvini, Ph.D, Study Chair — Universidade Federal de Sao Carlos
Locations (1):
- Industrial University of Santander UIS, Bucaramanga, Santander Department, Colombia

REFERENCES:
- [Background] Griffin JW, Newsome LS, Stralka SW, Wright PE. Reduction of chronic posttraumatic hand edema: a comparison of high voltage pulsed current, intermittent pneumatic compression, and placebo treatments. Phys Ther. 1990 May;70(5):279-86. doi: 10.1093/ptj/70.5.279. PMID 2185495
- [Background] Cosgrove KA, Alon G, Bell SF, Fischer SR, Fowler NR, Jones TL, Myaing JC, Crouse TM, Seaman LJ. The electrical effect of two commonly used clinical stimulators on traumatic edema in rats. Phys Ther. 1992 Mar;72(3):227-33. doi: 10.1093/ptj/72.3.227. PMID 1584856
- [Background] Taylor K, Mendel FC, Fish DR, Hard R, Burton HW. Effect of high-voltage pulsed current and alternating current on macromolecular leakage in hamster cheek pouch microcirculation. Phys Ther. 1997 Dec;77(12):1729-40. doi: 10.1093/ptj/77.12.1729. PMID 9413451
- [Background] Taylor K, Fish DR, Mendel FC, Burton HW. Effect of a single 30-minute treatment of high voltage pulsed current on edema formation in frog hind limbs. Phys Ther. 1992 Jan;72(1):63-8. doi: 10.1093/ptj/72.1.63. PMID 1728050
- [Background] Fish DR, Mendel FC, Schultz AM, Gottstein-Yerke LM. Effect of anodal high voltage pulsed current on edema formation in frog hind limbs. Phys Ther. 1991 Oct;71(10):724-30; discussion 730-3. doi: 10.1093/ptj/71.10.724. PMID 1946611
- [Background] Mendel FC, Wylegala JA, Fish DR. Influence of high voltage pulsed current on edema formation following impact injury in rats. Phys Ther. 1992 Sep;72(9):668-73. doi: 10.1093/ptj/72.9.668. PMID 1508974
- [Background] Bettany JA, Fish DR, Mendel FC. Influence of high voltage pulsed direct current on edema formation following impact injury. Phys Ther. 1990 Apr;70(4):219-24. doi: 10.1093/ptj/70.4.219. PMID 2315384
- [Background] Bettany JA, Fish DR, Mendel FC. High-voltage pulsed direct current: effect on edema formation after hyperflexion injury. Arch Phys Med Rehabil. 1990 Aug;71(9):677-81. PMID 2375674
- [Background] Karnes JL, Mendel FC, Fish DR. Effects of low voltage pulsed current on edema formation in frog hind limbs following impact injury. Phys Ther. 1992 Apr;72(4):273-8. doi: 10.1093/ptj/72.4.273. PMID 1584859
- [Background] Thornton RM, Mendel FC, Fish DR. Effects of electrical stimulation on edema formation in different strains of rats. Phys Ther. 1998 Apr;78(4):386-94. doi: 10.1093/ptj/78.4.386. PMID 9555921
- [Background] Dolan MG, Mychaskiw AM, Mendel FC. Cool-Water Immersion and High-Voltage Electric Stimulation Curb Edema Formation in Rats. J Athl Train. 2003 Sep;38(3):225-230. PMID 14608432
- [Background] Karnes JL, Mendel FC, Fish DR, Burton HW. High-voltage pulsed current: its influence on diameters of histamine-dilated arterioles in hamster cheek pouches. Arch Phys Med Rehabil. 1995 Apr;76(4):381-6. doi: 10.1016/s0003-9993(95)80665-2. PMID 7717840
- [Background] Dolan MG, Mychaskiw AM, Mattacola CG, Mendel FC. Effects of Cool-Water Immersion and High-Voltage Electric Stimulation for 3 Continuous Hours on Acute Edema in Rats. J Athl Train. 2003 Dec;38(4):325-329. PMID 14737215
- [Background] Dolan MG, Graves P, Nakazawa C, Delano T, Hutson A, Mendel FC. Effects of Ibuprofen and High-Voltage Electric Stimulation on Acute Edema Formation After Blunt Trauma to Limbs of Rats. J Athl Train. 2005 Jun;40(2):111-115. PMID 15970957
- [Background] Mohr TM, Akers TK, Landry RG. Effect of high voltage stimulation on edema reduction in the rat hind limb. Phys Ther. 1987 Nov;67(11):1703-7. doi: 10.1093/ptj/67.11.1703. PMID 3499622
- [Background] Cook HA, Morales M, La Rosa EM, Dean J, Donnelly MK, McHugh P, Otradovec A, Wright KS, Kula T, Tepper SH. Effects of electrical stimulation on lymphatic flow and limb volume in the rat. Phys Ther. 1994 Nov;74(11):1040-6. doi: 10.1093/ptj/74.11.1040. PMID 7972365
- [Background] Mendel FC, Fish DR. New Perspectives in Edema Control via Electrical Stimulation. J Athl Train. 1993 Spring;28(1):63-74. PMID 16558209
- [Background] Reed BV. Effect of high voltage pulsed electrical stimulation on microvascular permeability to plasma proteins. A possible mechanism in minimizing edema. Phys Ther. 1988 Apr;68(4):491-5. doi: 10.1093/ptj/68.4.491. PMID 2451258
- [Derived] Sandoval MC, Ramirez C, Camargo DM, Salvini TF. Effect of high-voltage pulsed current plus conventional treatment on acute ankle sprain. Rev Bras Fisioter. 2010 May-Jun;14(3):193-9. doi: 10.1590/s1413-35552010000300012. PMID 20730362
- See also: Universidad Industrial de Santander - Home page — http://www.uis.edu.co
- See also: Universidade Federal de Sao Carlos - Home page — http://www.ufscar.br